CLINICAL TRIAL: NCT00400608
Title: A Repeat-dose, Open-label, Randomized, Incomplete Block Design in Pediatric Subjects With Asthma, Ages 4 - 11 Years, to Compare Systemic Exposure and Pharmacodynamics of Fluticasone Propionate and Salmeterol Following Advair HFA 45/21mcg (2 Inhalations), ADVAIR® HFA 45/21mcg (2 Inhalations) With Aerochamber Plus Spacer and Advair Diskus 100/50 Twice Daily
Brief Title: A Study In Pediatric Subjects With Asthma Using ADVAIR HFA, ADVAIR HFA With Spacer, And ADVAIR DISKUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAS105519
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: pediatrics; ADVAIR Inhaler; Asthma; ADVAIR DISKUS
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ADVAIR HFA
Drug: ADVAIR DISKUS
  Other Names: ADVAIR HFA

SUMMARY:
Collect PK/PD data for this age group to compare ADVAIR DISKUS with ADVAIR HFA

DETAILED DESCRIPTION:
A repeat-dose open label randomized incomplete block design in pediatric subjects with asthma, ages 4-11 years, to compare systemic exposure and pharmacodynamics of fluticasone propionate and salmeterol following ADVAIR HFA 45/21mcg(2 inhalations), ADVAIR HFA 45/21mcg(2 inhalations) with Aerochamber Plus Spacer and ADVAIR DISKUS 100/50 twice daily

ELIGIBILITY:
Inclusion criteria:

* Subjects with mild asthma
* No significant medical conditions at screen
* Weigh at least 20 kg

Exclusion criteria:

* No clinical abnormalities at screen visit
* Asthma control at least 3 months prior with anti-steroidal medication only

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2006-10; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
PD of Fluticasone as measured by serum cortisol followed by doses of ADVAIR HFA and ADVAIR DISKUS | 3 Weeks

SECONDARY OUTCOMES:
To assess the exposure of FP and Salmeterol following the doses of ADVAIR HFA and ADVAIR DISKUS as well as assessing safety measurements based on adverse event reporting | 3 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Medford, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: SAS105519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SAS105519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SAS105519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SAS105519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SAS105519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SAS105519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SAS105519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register